CLINICAL TRIAL: NCT00481871
Title: A Phase 1/2a Open-label Study of Pralatrexate and Gemcitabine With Vitamin B12 and Folic Acid Supplementation in Patients With Relapsed or Refractory Lymphoproliferative Malignancies
Brief Title: Study of Pralatrexate & Gemcitabine With B12 & Folic Acid to Treat Relapsed/Refractory Lymphoproliferative Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Acrotech Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDX-009
Record Dates: First submitted 2007-06-01; First posted 2007-06-04 (Estimated); Results first posted 2012-09-18 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2019-12

CONDITIONS: Relapsed or Refractory Lymphoproliferative Malignancies; Hodgkin's Lymphoma; Peripheral T-cell Lymphoma; B-cell Lymphoma; Waldenstrom's Macroglobulinemia
Keywords: Lymphoproliferative malignancies; Lymphoma; Hodgkin's lymphoma (HL); Non-Hodgkin's lymphoma (NHL); PTCL; T/NK-cell leukemia/lymphoma; T-cell lymphoma/leukemia (HTLV 1+); Angioimmunoblastic T-cell lymphoma; Blastic NK lymphoma; Anaplastic large cell lymphoma; T/NK-cell lymphoma; Enteropathy-type intestinal lymphoma; Hepatosplenic T-cell lymphoma; Extranodal peripheral T/NK-cell lymphoma; Subcutaneous panniculitis T-cell lymphoma; Transformed mycosis fungoides; PDX; Pralatrexate; Gemcitabine; Gemzar; Vitamin B12; Folic acid
MeSH Terms: conditions — Recurrence; Hodgkin Disease; Lymphoma, T-Cell, Peripheral; Lymphoma, B-Cell; Waldenstrom Macroglobulinemia; Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, T-Cell; Leukemia; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Extranodal NK-T-Cell | interventions — 10-propargyl-10-deazaaminopterin; Gemcitabine; Commerce; WW Domain-Containing Oxidoreductase; Vitamin B 12; Folic Acid

ARMS (2):
- Pralatrexate & Gemcitabine - Sequential Days (Experimental)
  Interventions: Drug: Pralatrexate Injection; Drug: Gemcitabine Hydrochloride; Dietary Supplement: Vitamin B12; Dietary Supplement: Folic Acid
- Pralatrexate & Gemcitabine - Same Day (Experimental)
  Interventions: Drug: Pralatrexate Injection; Drug: Gemcitabine Hydrochloride; Dietary Supplement: Vitamin B12; Dietary Supplement: Folic Acid

INTERVENTIONS:
Drug: Pralatrexate Injection — Intravenous (IV) push administration over 30 seconds to 5 minutes into a patent IV line containing normal saline (0.9% sodium chloride).
  Sequential Dosing: 10 mg/m2 every 2 weeks (days 1 and 15) of a 4-week cycle until criteria for discontinuation per the protocol are met.
  Same Day Dosing: 15 mg/m2 every 2 weeks (days 1 and 15) of a 4-week cycle until criteria for discontinuation per the protocol are met.
  Other Names: FOLOTYN; PDX; Pralatrexate; (RS)-10-propargyl-10-deazaaminopterin
Drug: Gemcitabine Hydrochloride — Gemcitabine will be prepared and administered as an IV infusion as per manufacturer instructions.
  Sequential Dosing: 400 mg/m2 every 2 weeks (days 2 and 16) of a 4-week cycle until criteria for discontinuation per the protocol are met.
  Same Day Dosing: 600 mg/m2 every 2 weeks (days 1 and 15) of a 4-week cycle until criteria for discontinuation per the protocol are met.
  Other Names: Gemcitabine; Gemzar®, Eli Lilly and Company; Gemcitabine Hydrochloride (HCl) for Injection
Dietary Supplement: Vitamin B12 — 1 mg intramuscular injection
  Administered within 10 weeks of enrollment, every 8-10 weeks throughout the study and for at least 30 days after last dose of pralatrexate.
  Other Names: Cyanocobalamin
Dietary Supplement: Folic Acid — 1 mg orally
  Administered daily for at least 7 days prior to start of pralatrexate, throughout the study and for at least 30 days after last dose of pralatrexate.
  Other Names: Vitamin B9; Folate; Folacin

SUMMARY:
This study is for patients with lymphoproliferative malignancies that have progressed after receiving a previous treatment (relapsed) or are no longer responding to treatment (refractory). To be in this study, patients must have certain types of Hodgkin's lymphoma (HL), peripheral T-cell lymphoma (PTCL), or B-cell lymphoma, including Waldenstrom's macroglobulinemia.

This study is being done to find doses of the combination of pralatrexate and gemcitabine with vitamin B12 and folic acid that can be safely given to patients with these types of lymphoma and explore the effectiveness of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1: Histologically/cytologically confirmed lymphoproliferative malignancy. Patients with Hodgkin lymphoma (HL) or non-HL are eligible, with exceptions per exclusion criteria.
* Phase 2a: Histologically/cytologically confirmed HL, peripheral T-cell lymphoma (PTCL), or B-cell lymphoma including Waldenström's macroglobulinemia, with exceptions per exclusion criteria.
* Progression of disease (PD) after at least 1 prior treatment (any number of prior therapies allowed). PD after last prior treatment and recovered from toxic effects of prior therapy. Patients treated with an FDA-approved monoclonal antibody therapy may be enrolled at any time after the therapy if they have PD.
* PTCL patients must have received single-agent pralatrexate as a prior therapy.
* Eastern Cooperative Oncology Group performance status ≤ 2.
* Adequate blood, liver and kidney function per laboratory tests.
* Has taken 1 mg daily oral folic acid for at least 7 days prior to planned start of pralatrexate and received 1 mg vitamin B12 intramuscularly within 10 weeks of the planned start of pralatrexate.
* Females of childbearing potential must practice a medically acceptable contraceptive regimen from first dose until at least 30 days after last dose of pralatrexate and have a negative serum pregnancy test within 14 days prior to the first day of study treatment. Postmenopausal (defined as greater than 12 months since last menses) and surgically sterilized females do not require this test.
* Males who are not surgically sterile must practice a medically acceptable contraceptive regimen from first dose until at least 90 days after last dose of pralatrexate.
* Give written informed consent.

Exclusion Criteria:

* Phase 1

  1. B-cell: lymphoplasmacytic lymphoma (± Waldenström's macroglobulinemia); plasma cell myeloma/plasmacytoma; hairy cell leukemia.
* Phase 2a

  1. PTCL: precursor T/Natural Killer (NK) neoplasms, with the exception of blastic NK lymphoma; T-cell prolymphocytic leukemia; T-cell large granular lymphocytic leukemia; mycosis fungoides (MF), except transformed MF; Sézary syndrome; primary cutaneous CD30+ disorders: Anaplastic large cell lymphoma and lymphomatoid papulosis.
  2. B-cell: plasma cell myeloma/plasmacytoma; hairy cell leukemia.
* Relapsed HL or diffuse large B-cell lymphoma patients who are candidates for high dose therapy and autologous stem cell transplantation (SCT) and for whom it is a standard curative option.
* Active concurrent malignancy (except non melanoma skin cancer or carcinoma in situ of the cervix). If there is a history of prior malignancy, must be disease free for at least 5 years.
* Congestive heart failure Class III/IV.
* Uncontrolled hypertension.
* Human immunodeficiency virus (HIV)- positive diagnosis with CD4 less than 100 or detectable viral load within past 3 months and receiving anti-retroviral therapy.
* Hepatitis B or C virus with detectable viral load or immunological evidence of chronic active disease or receiving/requiring antiviral therapy.
* Central nervous system disease.
* Undergone an allogeneic SCT.
* Patients with disease refractory to peripheral blood SCT, or who have relapsed less than 100 days since an autologous or peripheral blood SCT.
* Active uncontrolled infection, underlying medical condition including unstable heart disease, or other serious illness impairing the ability to receive protocol treatment.
* Major surgery within 2 weeks of planned start of treatment.
* Receipt of any conventional chemotherapy or radiation therapy (encompassing greater than 10% of bone marrow) within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to study treatment or planned use during the study.
* Receipt of systemic corticosteroids within 7 days of study treatment, unless on a continuous dose of no more than 10 mg/day of prednisone for at least 1 month.
* Use of investigational drugs, biologics, or devices within 4 weeks prior to study treatment or planned use during the study.
* Received a monoclonal antibody within 3 months without evidence of PD.
* Previous exposure to pralatrexate and/or gemcitabine if discontinued due to treatment-related toxicity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2007-05; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Saunders, MD, Study Director — Spectrum Pharmaceuticals, Inc
Locations (15):
- United States (15):
  - University of California at Los Angeles, Los Angeles, California
  - Stanford University School of Medicine, Stanford, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - University of Chicago Hospital, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - The Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - New York University Hospital, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - UT MD Anderson Cancer Center, Houston, Texas
  - Cancer Therapy & Research Center, San Antonio, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between May 2007 and July 2010 across 16 study sites, all in the United States.
Pre-assignment Details: 12 patients were enrolled but not treated. Of these, 9 patients had events after enrollment that rendered them ineligible; 2 patients had progressive disease (PD); 1 patient withdrew consent. Since they were never dosed, these 12 patients were not included in efficacy or safety assessments.
Groups:
- Phase 1 Group A - Dose Finding: Phase 1 Treatment Group A had pralatrexate and gemcitabine administered on sequential days every week for 3 weeks followed by 1 week of rest (a 4 week cycle). The starting dose was 15 mg/m2 of pralatrexate and 400 mg/m2 of gemcitabine.
- Phase 1 Group B - Dose Finding: Phase 1 Treatment Group B had pralatrexate followed the next day by gemcitabine administered once every 2 weeks. One cycle of pralatrexate and gemcitabine was 4 weeks in duration and consisted of 2 doses each of pralatexate and gemcitabine. The starting dose was 10 mg/m2 of pralatrexate and 300 mg/m2 of gemcitabine.
- Phase 1 Group C - Dose Finding: Phase 1 Treatment Group C had pralatrexate followed 1 hour later by gemcitabine administered once every 2 weeks. One cycle of pralatrexate and gemcitabine was 4 weeks in duration and consisted of 2 doses each of pralatrexate and gemcitabine. The starting dose was 10 mg/m2 of pralatrexate and 300 mg/m2 of gemcitabine.
- Phase 2 Group B: Phase 2 Treatment Group B had 10 mg/m2 of pralatrexate followed the next day by 400 mg/m2 of gemcitabine administered once every 2 weeks. One cycle of pralatrexate and gemcitabine was 4 weeks in duration and consisted of 2 doses each of pralatexate and gemcitabine.
- Phase 2 Group C: Phase 2 Treatment Group C had 15 mg/m2 of pralatrexate followed 1 hour later by 600 mg/m2 of gemcitabine administered once every 2 weeks. One cycle of pralatrexate and gemcitabine was 4 weeks in duration and consisted of 2 doses each of pralatrexate and gemcitabine.
Period: Overall Study
Arm/Group | Phase 1 Group A - Dose Finding | Phase 1 Group B - Dose Finding | Phase 1 Group C - Dose Finding | Phase 2 Group B | Phase 2 Group C
Started | 7 | 10 | 18 | 38 | 34
Completed | 7 | 10 | 17 | 38 | 34
Not Completed | 0 | 0 | 1 | 0 | 0
Not completed — Progressive Disease - pt withdrew | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1 - Group A: Phase 1 Treatment Group A had pralatrexate and gemcitabine administered on sequential days every week for 3 weeks followed by 1 week of rest (a 4 week cycle). The starting dose was 15 mg/m2 of pralatrexate and 400 mg/m2 of gemcitabine.
- Phase 1 - Group B: Phase 1 Treatment Group B had pralatrexate followed the next day by gemcitabine administered once every 2 weeks. One cycle of pralatrexate and gemcitabine was 4 weeks in duration and consisted of 2 doses each of pralatexate and gemcitabine. The starting dose was 10 mg/m2 of pralatrexate and 300 mg/m2 of gemcitabine.
- Phase 1 - Group C: Phase 1 Treatment Group C had pralatrexate followed 1 hour later by gemcitabine administered once every 2 weeks. One cycle of pralatrexate and gemcitabine was 4 weeks in duration and consisted of 2 doses each of pralatrexate and gemcitabine. The starting dose was 10 mg/m2 of pralatrexate and 300 mg/m2 of gemcitabine.
- Phase 2 - Group B: Phase 2 Treatment Group B had 10 mg/m2 of pralatrexate followed the next day by 400 mg/m2 of gemcitabine administered once every 2 weeks. One cycle of pralatrexate and gemcitabine was 4 weeks in duration and consisted of 2 doses each of pralatexate and gemcitabine.
- Phase 2 - Group C: Phase 2 Treatment Group C had 15 mg/m2 of pralatrexate followed 1 hour later by 600 mg/m2 of gemcitabine administered once every 2 weeks. One cycle of pralatrexate and gemcitabine was 4 weeks in duration and consisted of 2 doses each of pralatrexate and gemcitabine.
- Total: Total of all reporting groups
Arm/Group | Phase 1 - Group A | Phase 1 - Group B | Phase 1 - Group C | Phase 2 - Group B | Phase 2 - Group C | Total
Number analyzed (Participants) | 7 | 10 | 18 | 38 | 34 | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 7 | 10 | 24 | 28 | 71
  >=65 years | 5 | 3 | 8 | 14 | 6 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (15) | 52.4 (18) | 57.4 (17) | 57.9 (16) | 53.2 (15) | 56.4 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 4 | 17 | 14 | 42
  Male | 3 | 7 | 14 | 21 | 20 | 65
Region of Enrollment [Number; unit: participants]
  United States | 7 | 10 | 18 | 38 | 34 | 107

OUTCOME MEASURES:

1. Primary Outcome: Objective Responses Assessed by International Workshop Criteria (IWC)
Description: Number of participants who achieved an objective response. Objective response was defined as a tumor response assessment of either complete response (CR) or partial response (PR) and was determined only for patients with measurable disease at baseline. A tumor response assessment reported by IWC without PET was used for any analyses in cases where an IWC+PET evaluation was not done.
Time Frame: Assessed every 8 weeks (+/- 1 week) for Phase II and no less than every 3 cycles for Phase I
Population: All patients who completed at least 1 cycle of treatment were included in the efficacy analysis
Measure: Number; unit: participants
Groups:
- Phase 1: Includes the Phase 1 dose-finding groups A, B, and C
Arm/Group | Phase 1 | Phase 2 - Group B | Phase 2 - Group C
Number analyzed (Participants) | 34 | 38 | 34
participants | 8 | 5 | 7

2. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the number of days between the date of first tumor response assessment of objective response to the time of the first tumor response assessment of progressive disease (PD) or death due to any cause (date of first PD assessment or death - date of first objective response assessment + 1)
Time Frame: Response assessments were performed no less than every 3 cycles in the Phase 1 part of the study and every 8 weeks (± 1 week) in the Phase 2a part of the study
Measure: Median (Full Range); unit: days
Arm/Group | Phase 1 | Phase 2 - Group B | Phase 2 - Group C
Number analyzed (Participants) | 8 | 5 | 7
days | 174 [35 to 288] | 210 [57 to 210] | 170 [59 to 178]

3. Secondary Outcome: Progression-free Survival (PFS) Time
Description: PFS time was calculated as the number of days from study day 1 to the date of PD or death, regardless of cause (date of PD or death - study day 1 + 1).
Time Frame: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 1 | Phase 2 - Group B | Phase 2 - Group C
Number analyzed (Participants) | 34 | 38 | 34
days | 53.0 [49.0 to 106.0] | 59.0 [52.0 to 99.0] | 54.0 [45.0 to 89.0]

ADVERSE EVENTS:
Groups:
- Phase 1: Patients that received at least one dose of pralatrexate in the Phase 1 portion of the study
Arm/Group | Phase 1 | Phase 2 - Group B | Phase 2 - Group C
Serious Adverse Events (participants affected / at risk) | 18/35 | 13/38 | 16/34
Other Adverse Events (participants affected / at risk) | 35/35 | 38/38 | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 (N=35) | Phase 2 - Group B (N=38) | Phase 2 - Group C (N=34)
altered state of consciousness (Nervous system disorders) | 1 | 0 | 0
arrhythmia (Cardiac disorders) | 1 | 0 | 0
cardiac failure congestive (Cardiac disorders) | 1 | 1 | 1
cellulitis (Infections and infestations) | 3 | 1 | 1
delirium tremens (Psychiatric disorders) | 1 | 0 | 0
febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 0
mental status changes (Psychiatric disorders) | 1 | 0 | 0
myocardial infarction (Cardiac disorders) | 2 | 0 | 0
pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
pneumonia (Infections and infestations) | 3 | 1 | 2
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
pyrexia (General disorders) | 2 | 4 | 7
tachycardia (Cardiac disorders) | 1 | 1 | 0
thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 1
thrombophlebitis superficial (Vascular disorders) | 1 | 0 | 0
upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
weight decreased (Investigations) | 1 | 0 | 0
sepsis (Infections and infestations) | 0 | 1 | 0
anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0
chills (General disorders) | 0 | 1 | 1
renal failure acute (Renal and urinary disorders) | 0 | 2 | 2
fatigue (General disorders) | 0 | 1 | 0
multi-organ failure (General disorders) | 0 | 1 | 0
bacteraemia (Infections and infestations) | 0 | 0 | 1
oral candidiasis (Infections and infestations) | 0 | 0 | 1
respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 1
sepsis syndrome (Infections and infestations) | 0 | 1 | 0
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2
atrial flutter (Cardiac disorders) | 0 | 0 | 1
bradycardia (Cardiac disorders) | 0 | 0 | 1
cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0
diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
stomatitis (Gastrointestinal disorders) | 0 | 0 | 2
hydronephrosis (Renal and urinary disorders) | 0 | 0 | 2
back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
hypotension (Vascular disorders) | 0 | 2 | 1
lymphoedema (Vascular disorders) | 0 | 1 | 0
femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2
cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0
rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
asthenia (General disorders) | 0 | 1 | 0
non-cardiac chest pain (General disorders) | 0 | 0 | 1
pain (General disorders) | 0 | 1 | 0
abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0
hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
ventricular arrhythmia (Cardiac disorders) | 0 | 1 | 0
urinary tract infection (Infections and infestations) | 0 | 0 | 1
accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
tumor lysis syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
pain management (Surgical and medical procedures) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 (N=35) | Phase 2 - Group B (N=38) | Phase 2 - Group C (N=34)
fatigue (General disorders) | 25 | 18 | 15
pyrexia (General disorders) | 23 | 18 | 15
chills (General disorders) | 6 | 12 | 4
oedema peripheral (General disorders) | 5 | 6 | 6
influenza like illness (General disorders) | 3 | 1 | 0
asthenia (General disorders) | 2 | 4 | 3
chest discomfort (General disorders) | 2 | 1 | 1
chest pain (General disorders) | 2 | 1 | 1
non-cardiac chest pain (General disorders) | 2 | 0 | 3
stomatitis (Gastrointestinal disorders) | 16 | 9 | 12
nausea (Gastrointestinal disorders) | 15 | 24 | 21
diarrhoea (Gastrointestinal disorders) | 13 | 11 | 8
vomiting (Gastrointestinal disorders) | 12 | 10 | 9
constipation (Gastrointestinal disorders) | 10 | 10 | 12
abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 4
abdominal pain (Gastrointestinal disorders) | 2 | 6 | 6
dysphagia (Gastrointestinal disorders) | 2 | 2 | 1
epigastric discomfort (Gastrointestinal disorders) | 2 | 0 | 1
gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 | 1
gingival pain (Gastrointestinal disorders) | 2 | 0 | 0
glossodynia (Gastrointestinal disorders) | 2 | 0 | 0
haematochezia (Gastrointestinal disorders) | 2 | 0 | 0
oral pain (Gastrointestinal disorders) | 2 | 3 | 2
anaemia (Blood and lymphatic system disorders) | 19 | 14 | 9
neutropenia (Blood and lymphatic system disorders) | 16 | 14 | 8
thrombocytopenia (Blood and lymphatic system disorders) | 14 | 16 | 8
leukopenia (Blood and lymphatic system disorders) | 5 | 4 | 3
febrile neutropenia (Blood and lymphatic system disorders) | 3 | 2 | 1
lymphopenia (Blood and lymphatic system disorders) | 2 | 1 | 0
pancytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 9
epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 2
cough (Respiratory, thoracic and mediastinal disorders) | 6 | 8 | 2
wheezing (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 1
hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 4
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 4
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1
dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
cellulitis (Infections and infestations) | 4 | 1 | 0
pneumonia (Infections and infestations) | 4 | 2 | 3
oral candidiasis (Infections and infestations) | 2 | 2 | 2
upper respiratory tract infection (Infections and infestations) | 2 | 3 | 3
dizziness (Nervous system disorders) | 8 | 5 | 8
paraesthesia (Nervous system disorders) | 8 | 0 | 1
headache (Nervous system disorders) | 7 | 9 | 6
neuropathy peripheral (Nervous system disorders) | 4 | 3 | 2
hypoaesthesia (Nervous system disorders) | 2 | 2 | 2
alanine aminotransferase increased (Investigations) | 4 | 3 | 4
alanine aminotransferase (Investigations) | 2 | 0 | 0
aspartate aminotransferase increased (Investigations) | 2 | 3 | 2
blood creatinine increased (Investigations) | 2 | 2 | 2
cardiac murmur (Investigations) | 2 | 0 | 0
platelet count decreased (Investigations) | 2 | 1 | 2
weight decreased (Investigations) | 2 | 0 | 1
white blood cell count (Investigations) | 2 | 0 | 0
rash (Skin and subcutaneous tissue disorders) | 5 | 2 | 2
alopecia (Skin and subcutaneous tissue disorders) | 4 | 2 | 0
pruritus (Skin and subcutaneous tissue disorders) | 4 | 5 | 5
erythema (Skin and subcutaneous tissue disorders) | 3 | 2 | 2
night sweats (Skin and subcutaneous tissue disorders) | 3 | 5 | 2
swelling face (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
back pain (Musculoskeletal and connective tissue disorders) | 5 | 4 | 3
muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0
neck pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 2
myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4
hypotension (Vascular disorders) | 6 | 3 | 3
flushing (Vascular disorders) | 2 | 1 | 2
hypertension (Vascular disorders) | 2 | 1 | 1
decreased appetite (Metabolism and nutrition disorders) | 5 | 3 | 1
anorexia (Metabolism and nutrition disorders) | 3 | 7 | 5
hyperuricaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
palpitations (Cardiac disorders) | 4 | 0 | 1
tachycardia (Cardiac disorders) | 3 | 3 | 2
myocardial infarction (Cardiac disorders) | 2 | 0 | 0
anxiety (Psychiatric disorders) | 3 | 3 | 1
abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 3
lip pain (Gastrointestinal disorders) | 0 | 2 | 0
pain (General disorders) | 1 | 2 | 4
memory impairment (Nervous system disorders) | 0 | 1 | 2
arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2
bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4 | 6
rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 7 | 1
rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
rales (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
neutrophil count decreased (Investigations) | 1 | 6 | 2
weight increased (Investigations) | 0 | 2 | 1
sepsis syndrome (Infections and infestations) | 0 | 2 | 0
dehydration (Metabolism and nutrition disorders) | 1 | 1 | 3
hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 5
hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 3
lacrimation increased (Eye disorders) | 0 | 1 | 2
renal failure acute (Renal and urinary disorders) | 0 | 2 | 3
ear pain (Ear and labyrinth disorders) | 0 | 3 | 1
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3
catheter site pain (General disorders) | 0 | 2 | 0
pitting oedema (General disorders) | 0 | 2 | 0
groin pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
dysgeusia (Nervous system disorders) | 0 | 2 | 1
urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
white blood cell count decreased (Investigations) | 1 | 3 | 1
blood lactate dehydrogenase increased (Investigations) | 0 | 2 | 0
sinus tachycardia (Cardiac disorders) | 0 | 1 | 2
bradycardia (Cardiac disorders) | 1 | 0 | 2
hydronephrosis (Renal and urinary disorders) | 1 | 0 | 2
incontinence (Renal and urinary disorders) | 0 | 2 | 0
insomnia (Psychiatric disorders) | 1 | 1 | 3
confusional state (Psychiatric disorders) | 0 | 1 | 2
vision blurred (Eye disorders) | 1 | 1 | 3
ocular hyperaemia (Eye disorders) | 1 | 0 | 2
urinary tract infection (Infections and infestations) | 3 | 1 | 2
haemoglobin decreased (Investigations) | 1 | 5 | 0
hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
hyponatraemia (Metabolism and nutrition disorders) | 1 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Allos agreements with investigators (PIs) may vary. The PI may publish/make public data from the trial after the earlier of publication by Allos or 18 months after study completion. Allos can review results communications prior to public release and can embargo communications regarding trial results for a period less than or equal to 90 days from submission for review. Allos can request changes to the communication related to confidential or patent information, or to ensure accuracy.